CLINICAL TRIAL: NCT02392598
Title: Effect of Hepatic Steatosis on Prognosis and Outcomes of Patients With Chronic Hepatitis B
Brief Title: A Hepatitis B With Hepatic Steatosis Study
Acronym: HBHS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fatty Liver and Alcoholic Liver Disease Study Group, China (Other)
Collaborators: Unimed Scientific Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HBV2015
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis B, Chronic; Hepatic Steatosis
MeSH Terms: conditions — Hepatitis B, Chronic; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an epidemiologic study on effect of hepatic steatosis on prognosis and outcomes of patients with chronic hepatitis B.

DETAILED DESCRIPTION:
This is a multicenter, prospective and open-enrollment epidemiologic study. All the patients with chronic hepatisis B will be enrolled in the study and followed up after 1 year, 3 years and 5 years with a visit window of +1 month.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed chronic hepatitis B.
2. Specific biopsy requirements for hepatic steatosis: qualified biopsy specimen within 6 months, >5% hepatocytes show macrovesicular steatosis under HE staining and X10 microscope.
3. Willing to participate in the long-term follow-up and cooperative.
4. Able to provide informed consent file.

Exclusion Criteria:

1. Unable to provide informed consent.
2. Patients are eligible for baseline analysis but not eligible for follow-up, if having any of the following condition:

   1. Any end-stage liver disease.
   2. Any malignant tumor.
   3. Any congenital liver disease such as Wilson disease.
   4. Any other serious disease of projected survival < 5 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients with chronic hepatisis B meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
liver cirrhosis | 5 years

SECONDARY OUTCOMES:
liver cancer | 5 years
liver failure | 5 years
type 2 diabetes | 5 years
cardiovascular and cerebrovascular events | 5 years
death | 5 years
response of hepatic steatosis to anti-virus treatment | 1 year
effect of hepatic steatosis on HBeAg negativation among patients without anti-virus treatment | 1 year
effect of hepatic steatosis on HBsAg negativation among patients without anti-virus treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiangao Fan, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (7):
- China (7):
  - Zhangzhou Zhengxing Hospital, Zhangzhou, Fujian
  - Shandong Provincial Hospital, Ji'nan, Shandong
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - Shanghai Xinhua Hospital, Shanghai